CLINICAL TRIAL: NCT05400772
Title: Does Core Activation on an Unstable Surface Affect Periscapular Muscle Activation?
Status: Unknown | Type: Observational
Last Known Status: Not yet recruiting
Sponsor: Hacettepe University (Other)
Responsible Party: Principal Investigator, Tuba Kaya Benli, lecturer, Hacettepe University
Other Study IDs: BAKİRCAYU
Record Dates: First submitted 2022-05-27; First posted 2022-06-02 (Actual); Last update posted 2022-06-02 (Actual); Status verified 2022-03

CONDITIONS: Healthy
Keywords: electromyography; muscle activation; exercise; scapula
MeSH Terms: conditions — Motor Activity

STUDY DESIGN:
Observational Model: Other | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Healthy subjects
  Interventions: Other: electromyographic device

INTERVENTIONS:
Other: electromyographic device — An 8-channel surface EMG system (Noraxon Telemyo DTS system, Scottsdale, USA) will be used to measure signals from muscles during surface electromyography measurements.

SUMMARY:
The core muscles contain various muscle groups that stabilize the shoulders, pelvis, and spine, and they play an important role as pivot points in extremity movements. It is known that core muscles stabilize the lumbar region and core stabilization affects muscle activation. İn addition conscious abdominal muscle activation during exercise performance is believed to promote greater scapular muscle activation through existing myofascial connections. Studies support the relationship between the scapular region and the core region.

Another aspect of rehabilitation is the use of unstable surfaces with exercise, since it is possible to increase neuromuscular demand without placing further overload on the musculoskeletal system.

Hypothesis originating from the investigation:

H1: Exercises performed with core activation on stable surfaces activate the muscles around the scapula more than exercises performed without core activation.

H2: Exercises performed with core activation on unstable surfaces activate the muscles around the scapula more than exercises performed without core activation.

H3: Exercises performed with core activation on unstable surfaces activate muscle activation around the scapula more than exercises performed on stable surfaces.

H4: Exercises performed without core activation on unstable surfaces activate muscle activation around the scapula more than exercises performed on stable surfaces.

DETAILED DESCRIPTION:
Muscle activation of upper trapezius, middle trapezius, lower trapezius ve serratus anterior will be measured by superficial electromyographic measurement. Muscle activation according to SENIAM for each muscle will be evaluated.

Muscle activations will be measured during 4 different scapula exercises based on the literature. These exercises are: Inferior glide, External rotation in sitting, External rotation with standing elevation, Wall slide.

The specified scapula exercises will be performed on stable and unstable surfaces while the core region muscles are active and inactive. During the exercises, superficial EMG measurements of muscles will be recorded bilaterally.

All measurements will be made in 3 repetitions.

ELIGIBILITY:
Inclusion Criteria:

* Young individuals aged 18 and over
* Body mass index <30kg/m2

Exclusion Criteria:

* Individuals with previous trauma, neurological or musculoskeletal disorders in the shoulder girdle, upper extremity, spine, or pelvic girdle
* Individuals with a limited or painful range of motion in the shoulder girdle, upper extremity, spine, or pelvic girdle

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: Young healthy individuals over the age of 18
Sampling Method: Non-Probability Sample
Enrollment: 30 (Estimated)
Dates: Start 2022-07-01 (Estimated); Primary Completion 2022-07-01 (Estimated); Study Completion 2022-09-01 (Estimated)

PRIMARY OUTCOMES:
Surface electromyographic measurement | 60 minutes
  Muscle activation measurement

CONTACTS AND LOCATIONS:
Overall Officials: Tuba KAYA BENLİ, Principal Investigator — İzmir Bakırçay University; Yeşim BAKAR, Prof., Study Director — İzmir Bakırçay University; Nuriye BÜYÜKTAŞ, Study Chair — İzmir Bakırçay University; Hüseyin MAHİROĞLU, Study Chair — İzmir Bakırçay University

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Barati A, Safarcherati A, Aghayari A, Azizi F, Abbasi H. Evaluation of Relationship between Trunk Muscle Endurance and Static Balance in Male Students. Asian J Sports Med. 2013 Dec;4(4):289-94. doi: 10.5812/asjsm.34250. Epub 2013 Nov 15. PMID 24800004
- [Background] Vega Toro AS, Cools AM, de Oliveira AS. Instruction and feedback for conscious contraction of the abdominal muscles increases the scapular muscles activation during shoulder exercises. Man Ther. 2016 Sep;25:11-8. doi: 10.1016/j.math.2016.05.331. Epub 2016 Jun 1. PMID 27422592
- [Background] de Oliveira Scatolin R, Hotta GH, Cools AM, Custodio GAP, de Oliveira AS. Effect of conscious abdominal contraction on the activation of periscapular muscles in individuals with subacromial pain syndrome. Clin Biomech (Bristol). 2021 Apr;84:105349. doi: 10.1016/j.clinbiomech.2021.105349. Epub 2021 Apr 2. PMID 33848705
- [Background] de Araujo RC, Nascimento VYS, Torres RJB, Trombini-Souza F, Behm D, Pitangui ACR. Can the Use of Unstable Surfaces and Instruction for Conscious Abdominal Contraction Increase the EMG Activity of the Periscapular Muscles During the Dynamic Push-Up? J Sport Rehabil. 2020 Feb 1;29(2):225-230. doi: 10.1123/jsr.2018-0165. PMID 30676180